CLINICAL TRIAL: NCT07319416
Title: Role of Dynamic Contrast-enhanced Ultrasound (D-CEUS) in Assessment of Response to Radioreceptor Therapy (PRRT) in Patients With Pancreatic and Gastrointestinal Tract Neuroendocrine Tumors (GEP-NET)
Brief Title: DCEUS to Assess Treatment Response to PRRT in GEP-NET
Acronym: DCEUS-PRRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof. Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7778
Record Dates: First submitted 2025-09-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: NET; Radionucleide Therapy; Contrast Enhanced Ultrasound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEP-NET (Experimental): NET patients enrolled who undergo CEUS in order to assess early treatment response to PRRT
  Interventions: Device: Vuebox

INTERVENTIONS:
Device: Vuebox — Software that analyses CEUS clips and derives time-intensity curves and quantitative numerical parameters that reflects contrast kinetic patterns.

SUMMARY:
Neuroendocrine tumors (NETs) are a wide group of neoplasms arising from the diffuse neuroendocrine cell system that features significant molecular and biological heterogeneity. They mainly derive from the enterochromaffin cells of the gastroenteropancreatic tract (GEP-NETs) and their incidence and prevalence are steadily rising, possibly as a consequence of improving diagnostic methods and earlier detection. A major feature of GEP-NETs is their somatostatin receptor (SSTR) immunogenicity, which is relevant both for diagnostic and therapeutic purposes.

For patients with unresectable or advanced disease, systemic treatment is the standard of care. In this setting, Somatostatin analogues (SSAs) are the standard first line therapy and, even if response rates are low, disease progression is halted in about two thirds of patient. Recently, targeted radionuclide therapy has claimed significant attention as a valuable treatment option for many solid neoplasms. This approach relies on the administration of a radionuclide linked to a carrier-molecule that selectively interacts with tumor associated antigens, being eventually internalized and releasing β-radiation emission and low-energy γ rays directly from the inside of the cancer cells. Peptide Receptor Radionuclide Therapy (PRRT) is strongly recommended in progressive metastatic/inoperable pretreated NETs that showed homogenous SSTRs expression by SSA positive PET-CT or single photon emission computed tomography (SPECT) imaging. Although PRRT is effective in the majority of cases, approximately 15-30% of patients will eventually progress during treatment. It is still challenging to distinguish potential responders versus non-responder patients. The identification of predictive biomarkers, apart from the required expression of somatostatin receptors, and of non-invasive diagnostic predictive exams, are an unmet need. Despite the promising clinical results, very little is known about the biological changes induced by PRRT on cancer tissue and tumor microenvironment and vascularization. The assessment of treatment' response therefore still relies on CT and PET-CT as markers of tumoral activity.

Among imaging modalities, ultrasound could play a key role in this setting. Indeed, contrast-enhanced ultrasound (CEUS) allows a thorough assessment of tumor perfusion through analysis of both contrast media flow pattern and time-intensity curves. This quantitative analysis, called dynamic contrast enhanced ultrasound (DCE-US) is a novel technique that estimates tissue perfusion based on phase-specific enhancement after the injection of microbubble contrast agents. The parameters derived from this analysis could be used for treatment monitoring in oncology, as they are easily comparable through time in each patient. In order to establish the bases for standardization of DCE-US, the European Federation of Societies for Ultrasound in Medicine and Biology (EFSUMB) recently published an update on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed diagnosis of unresectable, well-differentiated GEP-NET G2 or G3 according to WHO 2019 Classification with a Ki67 index > 2% up to 55%.
* Somatostatin receptor-positive (SSTR+) disease defined by a homogenous SSTRs expression by SSA positive PET-CT or SPECT imaging.
* At least one target lesion according to RECIST v1.1.
* Participants must have signed and dated an approved written informed consent and must be able to comply with any study specific procedure.

Exclusion Criteria:

* Known hypersensitivity to Lutetium 177Lu - radionuclides.
* Other known malignancies.
* Patients not able to declare meaningful informed consent on their own or any other vulnerable population to that.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tumour vascularization | - Firs evaluation: at baseline before initiation of PRRT - within 10 days after completion of any pre-planned PRRT therapy (which are planned every 8 weeks) - 6 months after last treatment - 9 months after last treatment
  • To evaluate the different patterns of tumor vascularization by dynamic contrast-enhanced ultrasound (DCE-US) at baseline, after completion of any pre-planned PRRT cycle and at post-treatment standard evaluation timepoint.
  DCE-US reports values of Echo-power in AU (arbitrary units) or time in seconds.
  Here's a list of quantitative features derived from DCE-US:
  * AT: Arrival time
  * FT: Fall time
  * MTT: Mean transit time
  * PE: Peak enhancement
  * TTP: Time to peak
  * WiAUC: Wash-in area under the curve
  * WiR: Wash-in rate
  * WiWoAUC: Wash-in and wash-out AUC
  * WoAUC: Wash-out AUC
  * WoR: Wash-out rate
  * RT: Rise time

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Universitario Agostino Gemelli, Rome, Rome, Italy